CLINICAL TRIAL: NCT02881164
Title: Effect of Glycemic Index of a Preparation on Postprandial Metabolic Parameters and Satiety in Subjects With Type 2 Diabetes Mellitus Under Intensive Insulin Therapy: Controlled Clinical Trial
Brief Title: Glycemic Index in Subjects With Diabetes Mellitus Insulin Requesting
Acronym: GIDMIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Principal Investigator, Claudia Vega Soto, Nutritionist, Universidad de Valparaiso
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-2015
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glycemia; Satiety; Insulin; Breakfast; Low glycemic index; High glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low glycemic index breakfast (Experimental): Low glycemic index breakfast (GI=45)
  Interventions: Other: Low glycemic index
- High glycemic index breakfast (Active Comparator): High glycemic index breakfast (GI=80)
  Interventions: Other: High glycemic index

INTERVENTIONS:
Other: Low glycemic index — Subjects intake a low glycemic index breakfast
  Arms: Low glycemic index breakfast
Other: High glycemic index — Subjects intake a high glycemic index breakfast
  Arms: High glycemic index breakfast

SUMMARY:
To evaluate the acute effect of a low and high glycemic index breakfast on the glycemic response and satiety in subjects with type 2 diabetes mellitus under intensive insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus diagnosis.
* Minimum period of six months under intensive insulin therapy.
* Fast insulin prescription before breakfast.
* 35 and 70 years of age.
* BMI between 25 and 39.9 Kg/m2.
* HbA1c less than or equal to 10 % (86mmol/mol)
* Menopausal women under hormone replacement therapy

Exclusion Criteria:

* Pregnant women.
* Puerperal women.
* Subjects with neurological disease, endocrine disorder no treatment, kidney disease in stage IV or V, cancer, liver disease, chronic obstructive pulmonary disease, human immunodeficiency virus.
* Subjects with history of stroke, acute myocardial infarction or gastrointestinal resection.

Ages: 47 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Glycemia | -15 up to 120 minutes
  Glycemia (mg/dL) to -15, 30, 60 and 120 minutes, with respect to breakfast intake
Satiety | Up to 120 minutes
  Visual Analog Scale (VAS) was applied immediate and tardy postprandial (two hours after eating breakfast).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lobos DR, Vicuna IA, Novik V, Vega CA. Effect of high and low glycemic index breakfast on postprandial metabolic parameters and satiety in subjects with type 2 diabetes mellitus under intensive insulin therapy: Controlled clinical trial. Clin Nutr ESPEN. 2017 Aug;20:12-16. doi: 10.1016/j.clnesp.2017.04.082. Epub 2017 May 11. PMID 29072163